CLINICAL TRIAL: NCT03818646
Title: Functional Respiratory Imaging During Pulmonary Exacerbations in Adults With Non-cystic Fibrosis Bronchiectasis
Brief Title: Functional Respiratory Imaging in Bronchiectasis
Acronym: FRIBE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: P02470
Record Dates: First submitted 2018-11-29; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Bronchiectasis
Keywords: Exacerbation; Functional respiratory imaging
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Functional Respiratory Imaging — Functional Respiratory Imaging (FRI) is a novel image based functional diagnostic tool that combines high-resolution CT scans (HRCT) at TLC and FRC with flow simulations (computational fluid dynamics - CFD) providing a 3D visualization and quantification of lung structure and function.

SUMMARY:
Four-week prospective single centre exploratory study in adults with bronchiectasis suffering a pulmonary exacerbation (defined as a change in one or more of the following: cough; sputum amount; sputum colour; breathlessness; fevers; and malaise).

The study will recruit ten adult subjects (male and female) who attend the Cambridge Centre for Lung Infection (CCLI) at the Royal Papworth Hospital, Cambridge, United Kingdom. The study will include individuals with a known diagnosis of bronchiectasis suffering a current pulmonary exacerbation. Participants seen during their usual clinic review with an exacerbation will be invited to participate and enrolled to commence the study that same day (day 0). Participants enrolled will undergo clinical review and a series of standard-of-care testing including sputum culture, lung function tests and blood analysis. Additional to these standard investigations, participants will also undertake a series of patient reported outcomes via validated respiratory questionnaires (Quality of Life - Bronchiectasis - QOL-B; & Leicester Cough Questionnaire - LCQ) and functional respiratory imaging (FRI). FRI consists of low dose high-resolution CT at full inspiration and expiration, combined with computational fluid dynamic testing.

Participants will be treated without delay according to standard of care treatment as per current international guidelines. Participants may be treated as either an inpatient or outpatient determined by the treating respiratory physician.

Follow up will occur on day 7, 14 and 28 post enrolment with serial CT imaging on days 0, 14 and 28. No scheduled follow up testing will be required beyond the day 28 visit, however all participants will receive a follow-up phone call at day 35.

The investigators hypothesize that changes in FRI parameters will be seen pre and post exacerbation treatment and will correlate with changes in lung function and patient reported outcomes. This will confirm FRI as a surrogate biomarker for assessing therapeutic response in future clinical trials in bronchiectasis.

DETAILED DESCRIPTION:
Four-week prospective single centre exploratory study in adults with bronchiectasis suffering a pulmonary exacerbation.

The study will endeavour to recruit ten adult subjects (male and female) who attend the Cambridge Centre for Lung Infection (CCLI) at the Royal Papworth Hospital, Cambridge, United Kingdom. The study will include individuals with a known diagnosis of bronchiectasis (defined as symptoms of chronic or recurrent bronchial infection with radiological evidence of abnormal and permanent dilation of bronchi) not from cystic fibrosis; and a current pulmonary exacerbation (defined as a 'deterioration in three or more of the following key symptoms for at least 48h: cough; sputum volume and/or consistency; sputum purulence; breathlessness and/or exercise tolerance; fatigue and/or malaise; haemoptysis AND that a clinician determines a change in bronchiectasis treatment is required).

In order to maximise subject recruitment and understanding of the study, all CCLI patients with bronchiectasis that are known to suffer frequent exacerbations (>2 per year) will be sent details of the trial including the Patient Information and Consent Form at the time of study commencement, prior to their individual enrolment. Subjects then seen during their usual clinic review with a pulmonary exacerbation will be invited to participate and enrolled to commence the study that same day (day 0). Participants enrolled will undergo clinical review and a series of standard testing including pulmonary function tests and blood analysis. Additional to these standard investigations, participants will also undertake a series of patient reported outcomes via validated respiratory questionnaires (Quality of Life - Bronchiectasis - QOL-B; & Leicester Cough Questionnaire - LCQ) and functional respiratory imaging (FRI). FRI consists of low dose high-resolution CT at total lung capacity (TLC) and functional residual capacity (FRC), combined with computational fluid dynamic testing (CFD).

Participants will be treated without delay according to standard usual care as per the current European Respiratory Society (ERS) and British Thoracic Society (BTS) Bronchiectasis Guidelines. Participants may be treated as either an inpatient or outpatient determined by the treating consultant respiratory physician.

Follow up will occur on day 7, 14 and 28 post enrolment. Participants will undergo clinical review and repeat testing according to the below schedule. No scheduled follow up testing will be required beyond the day 28 visit, however all participants will receive a follow up phone call at day 35.

Day 0: Initial consultation - presentation with a pulmonary exacerbation

* Recruitment, consent and enrolment
* History and clinical examination
* Bloods (WCC; neutrophil count; CRP)
* Pregnancy test (urine dipstick) - if appropriate
* Lung function testing (FEV1; FVC; TLC)
* Sputum collection
* Functional respiratory imaging (HRCT at TLC and FRC; may occur + 48 hours of enrolment)
* Patient reported outcomes / questionnaires (QOL-B; LCQ)
* Usual treatment commencement (as per current bronchiectasis guidelines)

Day 7: Mid-treatment follow up (as per usual standard of care)

* History and clinical review
* Bloods (WCC, neutrophil count; CRP)

Day 14: End of treatment follow up

* History and clinical examination
* Bloods (WCC; neutrophil count; CRP)
* Pregnancy test (urine dipstick) - if appropriate
* Lung function testing (FEV1; FVC; TLC)
* Functional respiratory imaging (HRCT at TLC and FRC; may occur +/- 48 hours of day 14)
* Patient reported outcomes / questionnaires (QOL-B; LCQ)

Day 28: Completion of study testing

* History and clinical examination
* Bloods (WCC; neutrophil count; CRP)
* Pregnancy test (urine dipstick) - if appropriate
* Lung function testing (FEV1; FVC; TLC)
* Functional respiratory imaging (HRCT at TLC and FRC; may occur +/- 48 hours of day 28)
* Patient reported outcomes (QOL-B; LCQ)

Day 35: Phone call by research team member

- No scheduled investigations

No scheduled follow up testing will be required beyond the day 28 visit other then a follow up phone call at day 35 (see above).

The investigators hypothesize that changes in FRI parameters will be seen pre and post exacerbation treatment and will correlate well with changes in lung function and patient reported outcomes. This will confirm FRI as a surrogate biomarker for assessing therapeutic response in future clinical trials in bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females ≥18 years and ≤ 80 years
* Current diagnosis of bronchiectasis (see above definition)
* Current pulmonary exacerbation (see above definition)

Exclusion Criteria:

* Severe obstructive airways disease (defined as FEV1 < 30%; FEV1/FVC < 70%)
* Diagnosis of other active chronic lung disease (asthma; ABPA; COPD; pulmonary fibrosis)
* Currently treated non-tuberculous mycobacterial disease
* Acute congestive cardiac failure
* Contra-indication or unable to perform HRCT imaging, including pregnancy
* Contra-indication or unable to perform pulmonary function testing
* Active lung malignancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will endeavour to recruit ten adult subjects (male and female) who attend the Cambridge Centre for Lung Infection (CCLI) at the Royal Papworth Hospital, Cambridge, United Kingdom. The study will include individuals with a known diagnosis of bronchiectasis (defined as symptoms of chronic or recurrent bronchial infection with radiological evidence of abnormal and permanent dilation of bronchi) not from cystic fibrosis; and a current pulmonary exacerbation (defined as a 'deterioration in three or more of the following key symptoms for at least 48h: cough; sputum volume and/or consistency; sputum purulence; breathlessness and/or exercise tolerance; fatigue and/or malaise; haemoptysis AND that a clinician determines a change in bronchiectasis treatment is required).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Airway volume | Days 0; 14; and 28
  Change in image based airway volume from FRI
Airway resistance | Days 0; 14; and 28
  Change in image based airway resistance from FRI
Lung volume | Days 0; 14; and 28
  Change in image based lung volume from FRI
Internal airflow distribution | Days 0; 14; and 28
  Change in image based internal airflow distribution from FRI
Airway wall thickness | Days 0;14; and 28
  Change in image based airway wall thickness from FRI
Blood vessel density | Days 0; 14; and 28
  Change in image based blood vessel density from FRI
Centreline evaluation (airway dimensions over distance into the lung). | Days 0; 14; and 28
  Change in image based centreline evaluation (airway dimensions over distance into the lung) from FRI

SECONDARY OUTCOMES:
Lung function | Days 0; 14; and 28
  Correlation of FRI to lung function (FEV1)
QOL-B | Days 0; 14; and 28
  Correlation of FRI to the QOL-B (Quality of Life Bronchiectasis) questionnaire
LCQ | Days 0; 14; and 28
  Correlation of FRI to the LCQ (Leicester Cough Questionnaire) questionnaire
CRP | Days 0; 14; and 28
  Correlation of FRI to CRP (C-reactive protein)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, MD, Study Director — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Hill AT, Haworth CS, Aliberti S, Barker A, Blasi F, Boersma W, Chalmers JD, De Soyza A, Dimakou K, Elborn JS, Feldman C, Flume P, Goeminne PC, Loebinger MR, Menendez R, Morgan L, Murris M, Polverino E, Quittner A, Ringshausen FC, Tino G, Torres A, Vendrell M, Welte T, Wilson R, Wong C, O'Donnell A, Aksamit T; EMBARC/BRR definitions working group. Pulmonary exacerbation in adults with bronchiectasis: a consensus definition for clinical research. Eur Respir J. 2017 Jun 8;49(6):1700051. doi: 10.1183/13993003.00051-2017. Print 2017 Jun. PMID 28596426
- [Background] Koser U, Hill A. What's new in the management of adult bronchiectasis? F1000Res. 2017 Apr 20;6:527. doi: 10.12688/f1000research.10613.1. eCollection 2017. PMID 28491293
- [Background] Quint JK, Millett ER, Joshi M, Navaratnam V, Thomas SL, Hurst JR, Smeeth L, Brown JS. Changes in the incidence, prevalence and mortality of bronchiectasis in the UK from 2004 to 2013: a population-based cohort study. Eur Respir J. 2016 Jan;47(1):186-93. doi: 10.1183/13993003.01033-2015. Epub 2015 Nov 5. PMID 26541539
- [Background] Chang AB, Bell SC, Byrnes CA, Grimwood K, Holmes PW, King PT, Kolbe J, Landau LI, Maguire GP, McDonald MI, Reid DW, Thien FC, Torzillo PJ. Chronic suppurative lung disease and bronchiectasis in children and adults in Australia and New Zealand. Med J Aust. 2010 Sep 20;193(6):356-65. doi: 10.5694/j.1326-5377.2010.tb03949.x. PMID 20854242
- [Background] Vendrell M, de Gracia J, Olveira C, Martinez-Garcia MA, Giron R, Maiz L, Canton R, Coll R, Escribano A, Sole A. [Diagnosis and treatment of bronchiectasis. Spanish Society of Pneumology and Thoracic Surgery]. Arch Bronconeumol. 2008 Nov;44(11):629-40. doi: 10.1157/13128330. Spanish. PMID 19007570
- [Background] Vos W, De Backer J, Poli G, De Volder A, Ghys L, Van Holsbeke C, Vinchurkar S, De Backer L, De Backer W. Novel functional imaging of changes in small airways of patients treated with extrafine beclomethasone/formoterol. Respiration. 2013;86(5):393-401. doi: 10.1159/000347120. Epub 2013 Apr 12. PMID 23595105
- [Background] De Backer LA, Vos W, De Backer J, Van Holsbeke C, Vinchurkar S, De Backer W. The acute effect of budesonide/formoterol in COPD: a multi-slice computed tomography and lung function study. Eur Respir J. 2012 Aug;40(2):298-305. doi: 10.1183/09031936.00072511. Epub 2011 Dec 19. PMID 22183484
- [Background] Hajian B, De Backer J, Vos W, Van Holsbeke C, Clukers J, De Backer W. Functional respiratory imaging (FRI) for optimizing therapy development and patient care. Expert Rev Respir Med. 2016 Feb;10(2):193-206. doi: 10.1586/17476348.2016.1136216. PMID 26731531
- [Background] van Geffen WH, Hajian B, Vos W, De Backer J, Cahn A, Usmani OS, Van Holsbeke C, Pistolesi M, Kerstjens HA, De Backer W. Functional respiratory imaging: heterogeneity of acute exacerbations of COPD. Int J Chron Obstruct Pulmon Dis. 2018 May 30;13:1783-1792. doi: 10.2147/COPD.S152463. eCollection 2018. PMID 29881268
- [Background] Bos AC, van Holsbeke C, de Backer JW, van Westreenen M, Janssens HM, Vos WG, Tiddens HA. Patient-specific modeling of regional antibiotic concentration levels in airways of patients with cystic fibrosis: are we dosing high enough? PLoS One. 2015 Mar 3;10(3):e0118454. doi: 10.1371/journal.pone.0118454. eCollection 2015. PMID 25734630